CLINICAL TRIAL: NCT04242238
Title: A Phase 1b Dose Escalation and Dose Expansion Study of a CSF1R Inhibitor (DCC-3014) Administered Concurrently With an Anti-PD-L1 Antibody (Avelumab) in Patients With Advanced High-grade Sarcoma
Brief Title: Study of DCC-3014 in Combination With Avelumab in Patients With Advanced or Metastatic Sarcomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: ENABLE MEDICINE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-340
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sarcoma; Advanced Sarcoma; High Grade Sarcoma; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma; Dedifferentiated Liposarcoma
Keywords: Advanced High Grade Sarcoma; CSF1R Inhibitor; DCC-3014; Anti-PD-L1 Antibody; Anti-PD-L1; Avelumab; Memorial Sloan Kettering Cancer Center; 19-340; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma; Dedifferentiated Liposarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Liposarcoma | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Standard 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced High-grade Sarcoma (Experimental): Dose Escalation: Up to 18 pts with locally advanced or metastatic high-grade sarcomas Dose Expansion: 10 pts per each diagnosis - undifferentiated pleomorphic sarcoma or myxofibrosarcoma, Leiomyosarcoma, Dedifferentiated liposarcoma
  Interventions: Drug: DCC-3014; Drug: Avelumab

INTERVENTIONS:
Drug: DCC-3014 — DCC-3014 will be administered in pill form. Start Day 1 on first cycle and continue with dosing of DCC-3014.
Drug: Avelumab — Start Day 1 on first cycle with further infusions of avelumab every 14 days

SUMMARY:
This study is being done to find the safest dose of DCC-3014 that can be given with avelumab to participants with advanced or metastatic sarcomas that will not cause serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years at the time of informed consent
* Be capable, willing, and able to provide written informed consent/assent
* Be willing to comply with clinical trial instructions and requirement, including mandatory biopsies
* Dose escalation phase: Patients must have a histologically confirmed metastatic and/or locally advanced high grade sarcoma
* Dose expansion phase: Patients must have a histologically confirmed metastatic and/or locally undifferentiated pleomorphic sarcoma, myxofibrosarcoma, leiomyosarcoma, or dedifferentiated liposarcoma
* Adequate performance status: ECOG 0 or 1/KPS 100-70%
* Patients must have at least one prior line of systemic therapy (e.g. chemotherapy, targeted or biological therapy) for their sarcoma. Prior neoadjuvant and/or adjuvant therapy will count regardless of when it was completed. Treatment naïve patients can enroll if they refuse standard of care systemic chemotherapy.
* Presence of measurable disease per RECIST v1.1. Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment
* Adequate organ function determined within 28 days of treatment initiation, as defined in Table 3:

Table 3: Laboratory values inclusion criteria

Hematological Absolute neutrophil count (ANC): ≥1,500 / mcL Platelets: ≥ 100,000 / mcL Hemoglobin: ≥ 9 g/dL or ≥ 5.6 mmol/L

Renal

Serum Creatinine OR Measured or calculated (Creatinine clearance should be calculated per institutional standard) creatinine clearance (GFR can also be used in place of creatinine or CrCl):

≤ 1.5 x upper limit of normal (ULN) OR ≥ 60 mL/min for patient with creatinine levels > 1.5 x institutional ULN

Hepatic Serum total bilirubin: ≤ 1.5 x ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT): ≤ 2.5 x ULN OR ≤ 5 x ULN for patient with liver metastases Albumin: ≥ 2.5mg/dL

Coagulation Internalized Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

* Women of childbearing potential (defined as a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months) must have a negative urine or serum pregnancy test at screening at ≤ 72 hours prior to day 1 of study treatment. If the urine pregnancy test if positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male and female patients of childbearing potential must be willing to use a highly effective method of contraception, for at least 30 days prior to the first dose of DCC-3014 and 7 months after the last dose of study medication. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient. Lactating w omen must be willing to not breastfeed during treatment and for at least one month after the last dose of Avelumab.

Exclusion Criteria:

* History of unstable or deteriorating cardiovascular disease within the previous 6 months prior to screening including but not limited to the following:

  * Unstable angina or myocardial infarction
  * CVA/stroke
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV)
  * Uncontrolled clinically significant arrhythmias
* Evidence or clinically significant interstitial lung disease or active, noninfectious pneumonitis related to prior immunotherapy treatment
* Malabsorption syndrome or other illness that could affect oral absorption
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases or carcinomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 day prior to trial treatment
* Current use of immunosuppressive medication, EXCEPT for the following:

  * intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses </= 10mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (>2 weeks) including oral steroid doses > 10mg/day of prednisone or equivalent within 2 months prior to enrollment
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease that is not controlled
* Patients known to be positive for active Hepatitis B (HBsAg reactive with detectable HBV DNA), or Hepatitis C (HCV RNA (qualitative) is detected)

  ° Patients with chronic hepatitis B (positive HBsAg and/or HBcAb and negative HBV DNA by PCR) are eligible for this study if deemed safe by a gastroenterologist
* Prolonged QTcF > 450 ms for men and >470 ms for women at Screening
* Patients who have received a live vaccine within 30 days of the start date of the planned study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Has a known history of active TB (Bacillus Tuberculosis)
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Alopecia, neuropathy Grade </= 2, or other Grade </= not constituting a safety risk based on investigator's judgment are acceptable
  * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy events due to a previously administered agent
* Patients who have received prior treatment with an anti-PD-1/PD-L1 agent
* Women who are pregnant or breast feeding
* Patients expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment(s)
* Prior organ transplantation including allogenic stem-cell transplantation
* Active infection requiring systemic therapy
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade >/= 3)
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  Identify the maximum tolerated dose (MTD) by evaluating toxicity using NCI CTCAE (version 4.03)
Overall Response Rate | 48 weeks
  Best overall response rate (CR+PR) based on RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org